CLINICAL TRIAL: NCT05008809
Title: Post-resection/Ablation Chemotherapy in Patients With Metastatic Colorectal Cancer Prospective, Randomized, Open, Multicenter Phase III Trial to Investigate the Efficacy of Active Post-resection/Ablation Therapy in Patients With Metastatic Colorectal Cancer
Brief Title: Post-resection/Ablation Chemotherapy in Patients With Metastatic Colorectal Cancer (FIRE-9 - PORT / AIO-KRK-0418)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dominik Paul Modest (Other)
Collaborators: German Research Foundation (Other); Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor-Investigator, Dominik Paul Modest, Prof. Dr. med., Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIRE-9 - PORT; AIO-KRK-0418 (Other: AIO); 2020-006144-18 (EudraCT Number)
Record Dates: First submitted 2021-08-06; First posted 2021-08-17 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Leucovorin; Oxaliplatin; Fluorouracil; Irinotecan; IFL protocol

STUDY DESIGN:
Intervention Model Description: open-label, randomized, controlled, multicenter, phase III study with two parallel arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Active treatment with mFOLFOXIRI or mFOLFOX6 or FOLFIRI q2w or CAPOX q3w up to six months followed by structured Follow-up for up to five years after randomization
  Interventions: Drug: mFOLFOX6; Drug: mFOLFOXIRI; Drug: FOLFIRI; Drug: CAPOX
- Control (No Intervention): Structured Follow-up for up to five years after randomization

INTERVENTIONS:
Drug: mFOLFOX6 — Oxaliplatin: 85 mg/m², 2h IV infusion on d1 Folinic acid: 400 mg/m², 1-2 h IV infusion on d1 5-FU: (optional: 400 mg/m² bolus, 2-5 min IV infusion), 2400 mg/m², 46 h IV infusion on d1 Cycles are repeated on day 15. A total of up to 12 cycles are administered.
  Other Names: Folinic acid, Oxaliplatin, 5-fluorouracil (FU)
  Arms: Treatment
Drug: mFOLFOXIRI — Oxaliplatin: 85 mg/m², 2h IV infusion on d1 Irinotecan: 150 mg/m², 90 min IV infusion on d1 Folinic acid: 400 mg/m², 1-2 h IV infusion on d1 5-FU: 2400 mg/m², 46 h IV infusion on d1 Cycles are repeated on day 15. A total of up to 12 cycles are administered.
  Other Names: Folinic acid, Oxaliplatin, 5-FU, Irinotecan
  Arms: Treatment
Drug: FOLFIRI — Folinic acid: 400mg/m², 1-2h IV Infusion on d1 5-FU: 2400 mg/m², 46 h IV infusion on d1 Irinotecan: 180 mg/m², 90-120 min IV infusion on d1 Cycles are repeated on day 15. A total of up to 12 cycles is administered.
  Other Names: Folinic acid, 5-FU
  Arms: Treatment
Drug: CAPOX — Capecitabine: 1000 mg/m², oral 1-0-1 on d1-14 Oxaliplatin: 130 mg/m², 3h IV infusion on d1 Cycles are repeated on day 22. A total of up to 8 cycles isadministered.
  Other Names: Capecitaine, Oxaliplatin
  Arms: Treatment

SUMMARY:
This is an open-label, randomized, controlled, multicenter, phase III study with two parallel arms. Patients with metastatic colorectal cancer after definite interventional therapy of all lesions are randomized in a 2:1 fashion (favoring active therapy) to investigate the efficacy, patient reported quality of life and safety of mFOLFOXIRI/mFOLFOX-6 as additive treatment (Arm A) versus active follow-up/surveillance (Arm B).

DETAILED DESCRIPTION:
The trial will consist of both a clinical and translational part. During the study, re-assessments (radiologic assessment, blood and QoL) will be conducted for all trial subject of the trial every 3 months. Tumor biopsies will be collected at screening (baseline sample) and in case of relapse of disease if a new tumor sample is obtained.

The objective of the re-assessments is detection of relapse either radiologically or within the translational material (blood samples with ctDNA dynamics and tumor - if available from relapses). CT scans of thorax/abdomen and/or MRI scans will be performed every 3 months within the 2 years after randomization. After the first two relapse-free years, intervals should be stretched to 6 months in the third and following years after study start. Structured follow-up for up to 60 months after randomization should be maintained for both arms.

Patients in Arm A receive additive study drug intervention (mFOLFOXIRI or mFOLFOX-6) for up to six months (12 cycles) after randomization with additional clinical and safety assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's signed informed consent.
2. Patient's age ≥18 years at the time of signing the informed consent.
3. Histologically confirmed adenocarcinoma of the colon or rectum.
4. Resected (R0 or R1) and/or effectively treated metastases (all techniques allowed) of colorectal cancer within 3-10 weeks before randomization (earlier randomisation allowed if at least 3 weeks interval between intervention and treatment start is guaranteed) AND resected primary tumor (synchronous or metachronous). In cases of synchronous metastases the interval of 3-10 weeks might be calculated following the removal of the primary tumor if this intervention was the last to address all tumor lesions.
5. Absence of significant active wound healing complications (if applicable) at randomization. Resolved wound healing complications after resection/ablation are acceptable for inclusion into the trial.
6. No radiographic evidence of active metastatic disease at study entry in a CT and/or MRI scan not older than 10 weeks prior randomization. Pre-surgery/ablation images are eligible for the study if all lesions have been addressed in the interval.
7. ECOG performance status 0-2.
8. Adequate bone marrow, hepatic and renal organ function, defined by the following laboratory test results:

   * Absolute neutrophil count >= 1.5 x 109/L (1500/µL)
   * Hemoglobin ≥ 80 g/L (8 g/dL)
   * Platelet count ≥ 100 x109/L (100000/µL) without transfusion
   * Total serum bilirubin of ≤ 1.5 x upper limit of normal (ULN)
   * Aspartate aminotransferase (AST/GOT) ≤ 3.0 × ULN.
   * Calculated glomerular filtration rate (GFR) according to Cockcroft-Gault formula or according to MDRD ≥ 50 mL/min or serum creatinine ≤ 1.5 x ULN
9. Patients without anticoagulation need to present with an INR < 1.5 x ULN and PTT < 1.5 x ULN. Patient with prophylactic or therapeutic anticoagulation are allowed into the trial.
10. Proficient fluorouracil metabolism as defined:

    1. Prior treatment with 5-FU or capecitabine without unusual toxicity or
    2. If tested, normal DPD deficiency test according to the standard of the study site or
    3. If tested, in patients with DPD deficiency test with a CPIC activity score of 1.0-1.5 fluoropyrimidine/capecitabine dosage should be reduced by 50%
11. For women of childbearing potential (WOCBP): negative pregnancy test within 14 days before randomization and agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for at least 9 months after the last dose of Oxaliplatin or for at least 6 months after the last dose of all other study treatment.

A woman is considered to be of childbearing potential if she is post-menarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male partner's sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

For men: With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for 6 months after the last dose of study treatment. Men must refrain from donating sperm during this same period.

Exclusion Criteria:

1. Treatment of metastases greater than 3 cm with radio-frequency/microwave ablation within 24 months prior to study entry if applicable.
2. Treatment of metastases greater than 5 cm with radiation (stereotactic/ brachytherapy) within 24 months prior to study entry if applicable.
3. Any previous systemic therapy is allowed for inclusion into the trial. However, if previous oxaliplatin-containing chemotherapy at any time for metastatic or localized disease was carried out, the inclusion into the trial is permitted under the condition, that

   1. A total duration of oxaliplatin-based therapy of six months (i.e. 12 cycles of FOLFOX / FOLFOXIRI or 8 cycles CAPOX) is not exceeded - including therapy within the FIRE-9/PORT trial
   2. If already more than three months of oxaliplatin-based therapy (i.e. >6 cycles of FOLFOX / FOLFOXIRI or >4 cycles CAPOX) was used, the study therapy should be started with an irinotecan-based regimen (i.e. FOLFIRI or FOLFOXIRI) However, in the case of FOLFOXIRI therapy in the trial, the above mention regulation concerning the total dosing of oxaliplatin still applies (i.e. 12 cycles of FOLFOX / FOLFOXIRI or 8 cycles CAPOX should not be exceeded - including therapy within the FIRE-9/PORT trial).
4. New York Heart Association Class III or greater heart failure by clinical judgement.
5. Myocardial infarction within 6 months prior to randomization; percutaneous transluminal coronary angioplasty (PTCA) with or without stenting within 6 months prior to randomization.
6. Unstable angina pectoris.
7. Unstable cardiac arrhythmia > grade 2 NCI CTCAE despite anti-arrhythmic therapy.
8. Ongoing toxicities > grade 2 NCI CTCAE
9. Active uncontrolled infection by investigator's perspective.
10. Severe chronic non-healing wounds, ulcerous lesions or untreated bone fracture.
11. Known hypersensitivity to 5-FU, folinic acid, irinotecan, oxaliplatin or capecitabine or to any of the other excipients listed in section 6.1 of the corresponding SmPC.
12. Recent or concomitant treatment with brivudine.
13. Peripheral sensitive neuropathy with functional impairment (> grade 1 acc. to CTCAE version 5.0 (see appendix 2)).
14. Inflammatory bowel disease and/or bowel obstruction.
15. Simultaneous application of Johannis herbs preparations.
16. Pernicious or other megaloblastic anemia caused by vitamin B12 deficiency.
17. Major surgical procedure, open biopsy, or significant traumatic injury within 21 days prior to randomization or at least to intended treatment start, or anticipation of need for major surgical procedure during the course of the study or non-recovery from side effects of any such procedure.
18. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications.
19. Medical history of malignant disease other than mCRC with the following exceptions:

    * patients who have been disease-free for at least three years before randomization
    * patients with adequately treated and completely resected basal cell or squamous cell skin cancer, in situ cervical, breast or prostate cancer, stage I uterine cancer
    * patients with any treated or untreated malignant disease that is associated with a 5-year survival prognosis of ≥ 90% and does not require active therapy
20. Known alcohol or drug abuse.
21. Pregnant or breastfeeding females.
22. Participation in a clinical trial or experimental drug treatment within 28 days prior to potential inclusion in the clinical trial or within a period of 5 half-lives of the substances administered in a clinical trial or during an experimental drug treatment prior to potential inclusion in the clinical trial, depending on which period is longest, or simultaneous participation in another clinical trial while taking part in this clinical trial.
23. Patients depending on Sponsor, investigator or study site.
24. Suspected SARS-CoV-2 infection with or without symptoms (evaluation according to local policy in respective center with respect to actual status of pandemic and with reference to the policy that would apply to patients with similar therapy outside the trial). This may include assessment of vaccination status, anamnesis, physical examination and potentially antigen and/or PCR testing.
25. Patient committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.
26. Limited legal capacity.
27. Concomitant administration of strong CYP3A4 and/or UGT1A1 inducers (e.g. Rifampicin, Carbamazepin, Phenobarbital, Phenytoin or Apalutamid).
28. Planned inoculation/vaccination with a live vaccine during treatment with Oxaliplatin and/or Irinotecan, and until 6 months after treatment with Irinotecan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) time | 24 months
  time from randomization to death or evidence of disease relapse/progression (whatever occurs first)

SECONDARY OUTCOMES:
Overall survival (OS) | at least 5 years after randomization
  time from randomization to the date of death of any cause
Control ol lesions | up to 5 years after randomization
  Local or distant control of lesions according to ablative technique (surgery vs. ablation vs. radiation)
(Serious) Adverse Events | up to 2 years after randomization
  Type, incidence, severity, and causal relationship to active chemotherapy of non-serious adverse events and serious adverse events (severity evaluated according to CTCAE version 5.0)
Quality of life (QoL) | up to 5 years after randomization
  Quality of life (QoL) as assessed with the QoL questionnaire EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Modest, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (79):
- Germany (79):
  - Klinikum St. Marien Amberg, Amberg
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Klinikum Bayreuth, Bayreuth
  - Charité Universitätsmedizin Berlin, Berlin
  - Helios Klinikum Emil von Behring, Berlin
  - MVZ Onkologischer Schwerpunkt am Oskar-Helene-Heim, Berlin
  - Vivantes Klinikum am Urban Berlin, Berlin
  - Vivantes Klinikum Spandau Berlin, Berlin
  - St. Josef-Hospital Bochum, Bochum
  - Johanniterkrankenhaus Bonn, Bonn
  - Diakonie-Krankenhaus Bremen, Bremen
  - Klinikum Chemnitz, Chemnitz
  - Kliniken der Satdt Köln, Cologne
  - Klinikum Darmstadt, Darmstadt
  - DONAUISAR Klinikum Deggendorf, Deggendorf
  - Städtisches Klinikum Dessau, Dessau
  - Onkologische-Gemeinschaftspraxis Dresden, Dresden
  - Onkozentrum Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Kliniken Essen-Mitte, Essen
  - Universitätsklinikum Essen, Essen
  - KHNW Frankfurt, Frankfurt
  - Markus-Krankenhaus Frankfurt, Frankfurt
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Gemeinschaftspraxis internistische Onkologie Fürth, Fürth
  - Niels-Stensen Kliniken Georgsmarienhütte, Georgsmarienhütte
  - Praxis Hämatologie Onkologie Gießen, Giessen
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Halle, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - St. Anna Hospital Herne, Herne
  - Universitätsklinikum des Saarlandes, Homburg
  - Klinikum Ingolstadt GmbH, Ingolstadt
  - Universitätsklinikum Jena, Jena
  - Klinikum Landshut, Landshut
  - VK&K Studien Landshut, Landshut
  - Studienzentrum UnterEms Leer, Leer
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum Leverkusen, Leverkusen
  - Klinikum Lippe, Lippe
  - Klinikum Ludwigsburg, Ludwigsburg
  - Klinikum Magdeburg, Magdeburg
  - Universitätsmedizin Mainz, Mainz
  - OnkoNet Marburg GmbH, Marburg
  - Philipps-Universität Marburg, Marburg
  - Johannes Wesling Klinikum Minden, Minden
  - Kliniken Maria Hilf Mönchengladbach, Mönchengladbach
  - Klinikum der Universität München, München
  - Klinikum rechts der Isar TU München, München
  - München Klinik Bogenhausen, München
  - München Klinik Neuperlach, München
  - Gemeinschaftspraxis Münster, Münster
  - Universitätsklinikum Münster, Münster
  - Friedrich-Ebert-Krankenhaus Neumünster, Neumünster
  - Lukaskrankenhaus Neuss, Neuss
  - Klinikum Nürnberg, Nuremberg
  - Pi.Tri-Studien GmbH Offenburg, Offenburg
  - Klinikum Passau, Passau
  - Schwerpunktpraxis Penzberg, Penzberg
  - Ernst von Bergmann Klinikum Potsdam, Potsdam
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - Krankenhaus Barmherzige Brüder Regensburg, Regensburg
  - Universitätsklinikum Regensburg, Regensburg
  - Kreiskliniken Reutlingen, Reutlingen
  - Mathias Spital Rheine, Rheine
  - RoMed Klinikum Rosenheim, Rosenheim
  - Universitätsmedizin Rostock, Rostock
  - DIAK Klinikum Schwäbisch Hall, Schwäbisch Hall
  - Marienkrankenhaus Siegen, Siegen
  - Klinikum Stuttgart, Stuttgart
  - Marienhospital Stuttgart, Stuttgart
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Universitätsklinikum Ulm, Ulm
  - Klinikum Wetzlar, Wetzlar
  - Onkologisches Zentrum Wolfsburg-Helmstedt, Wolfsburg
  - Petrus-Krankenhaus Wuppertal, Wuppertal
  - Gemeinschaftspraxis Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raschzok N, Stintzing S, Heinemann V, Rauch G, Ricke J, Guckenberger M, Kurreck A, Alig AHS, Stahler A, Bullinger L, Schmelzle M, Schoning W, Lurje G, Krenzien F, Haase O, Rau B, Gebauer B, Sauer IM, Pratschke J, Modest DP. FIRE-9 - PORT / AIO-KRK-0418: a prospective, randomized, open, multicenter Phase III trial to investigate the efficacy of adjuvant/additive chemotherapy in patients with definitely-treated metastatic colorectal cancer. BMC Cancer. 2022 Apr 2;22(1):359. doi: 10.1186/s12885-022-09422-6. PMID 35366831

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT05008809/Prot_SAP_000.pdf